CLINICAL TRIAL: NCT00282867
Title: Glucose Regulation in Acute Stroke Patients (GRASP) Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Karen C. Johnston, MD, MSc, PI, Professor and Chair Department of Neurology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11901; R01NS050192 (NIH)
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Results first posted 2009-08-21 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-07

CONDITIONS: Stroke; Hyperglycemia
Keywords: stroke; acute ischemic stroke; hyperglycemia; glucose; insulin; insulin and potassium therapy; GIK
MeSH Terms: conditions — Stroke; Hyperglycemia; Ischemic Stroke; Insulin Resistance | interventions — Potassium; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- tight control group (Active Comparator): target glucose level 70-110 mg/dL
  Interventions: Drug: IV glucose insulin and potassium, GIK
- loose control group (Active Comparator): target glucose level 70 - 200 mg/dL
  Interventions: Drug: IV glucose insulin and potassium, GIK
- usual care group (Active Comparator): target level 70 - 300 mg/dL
  Interventions: Other: standard care

INTERVENTIONS:
Drug: IV glucose insulin and potassium, GIK — The treatment intervention includes glucose, insulin, potassium infusion or standard therapy.
  Arms: loose control group; tight control group
Other: standard care — usual care
  Arms: usual care group

SUMMARY:
The purpose of this study is to assess the feasibility, safety and preliminary efficacy of the use of insulin infusions as treatment for hyperglycemic acute ischemic stroke patients.

DETAILED DESCRIPTION:
Ischemic stroke is a common, devastating and costly disease. Half of acute stroke patients have elevated glucose levels upon admission to the hospital, and hyperglycemia is associated with poor outcome for post-stroke patients. It is unclear if treatment of hyperglycemia or glucose lowering improves outcome, however, in animal stroke models and other human conditions, aggressive glucose lowering is beneficial.

The goal of this multicenter trial is to determine if tight control of blood glucose is beneficial in hyperglycemic patients with acute ischemic stroke. In the trial, researchers will compare intravenous (IV) glucose insulin and potassium (GIK) therapy plus meal insulin to control therapy in 72 stroke patients.

Participants will be randomly assigned to one of three groups-(1) the control group with a target glucose level of <300mg/dL; (2) the tight control GIK plus meal insulin group with a target of <110mg/dL; or (3) the loose control GIK plus meal insulin group with a target of <200mg/dL-with all groups avoiding glucose levels of <70mg/dL.

The specific aims of this study are to collect preliminary data on the safety and feasibility of GIK for treatment of hyperglycemia in acute stroke patients, and to collect preliminary data comparing tight GIK therapy with loose GIK therapy and control therapy. Information learned in this study will compliment ongoing work and allow for maximum efficiency in the design of future treatment trials.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Clinical diagnosis of ischemic stroke defined as acute neurological deficit occurring in one or more major vessels.
* Must arrive at hospital and be able to begin treatment within 2 hours of established eligibility and this must be within 24 hours of symptom onset. - - Patients unable to report symptom onset time or those awakening with symptoms must use the time last known to be well as the onset time.
* Admission plasma glucose of > 110 mg/dL.

Exclusion Criteria:

* Renal dysfunction as defined by a serum creatinine of >/=2.5 mg/dL at enrollment.
* Substantial pre-existing neurological or psychiatric illness that would confound neurological assessment.
* Patients who have received experimental therapy for the enrollment stroke.
* Pregnant females.
* Patients with other severe life threatening conditions that makes them unlikely to survive 90 days.
* Patients who are unable to follow the protocol or come back for 90-day followup.
* Patient has condition for which insulin infusion is the usual practice or the treating physician feels that there is an indication for insulin infusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2006-05; Primary Completion 2008-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Johnston, MD, Principal Investigator — University of Virginia, Department of Neurology
Locations (2):
- United States (2):
  - Medical College of Georgia, Augusta, Georgia
  - University of Virginia, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tight Control Group | Loose Control Group | Usual Care Group
Started | 24 | 25 | 25
Completed | 23 | 24 | 25
Not Completed | 1 | 1 | 0
Not completed — d/c prior to prim outcome, 3 m f/u done | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tight Control Group | Loose Control Group | Usual Care Group | Total
Number analyzed (Participants) | 24 | 25 | 25 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 8 | 12 | 31
  >=65 years | 13 | 17 | 13 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 10 | 33
  Male | 13 | 13 | 15 | 41
Region of Enrollment [Number; unit: participants]
  United States | 24 | 25 | 25 | 74

OUTCOME MEASURES:

1. Secondary Outcome: Favorable 3 Month Modified Rankin
Description: 3 month functional outcomes by modified Rankin (0 to 1) dichotomized as favorable versus not favorable outcome. Construct is functional handicap.
Time Frame: 3 months
Measure: Number; unit: percentage of participants
Arm/Group | Tight Control Group | Loose Control Group | Usual Care Group
Number analyzed (Participants) | 23 | 24 | 25
percentage of participants | 42 | 25 | 33

2. Primary Outcome: Hypoglycemic Events
Description: hypoglycemic events
Time Frame: up to 5 days
Measure: Number; unit: participants
Arm/Group | Tight Control Group | Loose Control Group | Usual Care Group
Number analyzed (Participants) | 23 | 24 | 25
participants | 7 | 1 | 1

3. Other Pre Specified Outcome: Symptomatic Hypoglycemia
Description: symptomatic hypoglycemia (glucose < 55 mg/dL)during treatment period
Time Frame: up to 5 days
Measure: Number; unit: participants
Arm/Group | Tight Control Group | Loose Control Group | Usual Care Group
Number analyzed (Participants) | 23 | 24 | 25
participants | 0 | 1 | 0

4. Post Hoc Outcome: Target Glucose Concentration
Description: glucose in target range in first 24 hours
Time Frame: first 24 hours after initiation of treatment
Population: Per protocol no analysis of this endpoint was performed in the "usual care" group.
Measure: Number; unit: participants
Arm/Group | Tight Control Group | Loose Control Group | Usual Care Group
Number analyzed (Participants) | 23 | 24 | 0
participants | 10 | 22 |

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No